CLINICAL TRIAL: NCT03895814
Title: Protective Step Training in People With Parkinson's Disease and Postural Disturbances
Brief Title: Protective Step Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Utah (Other); Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008325
Record Dates: First submitted 2019-03-19; First posted 2019-03-29 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease
Keywords: Balance; Falls; Posture; Cognition; Training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Multi-baseline assessment
Masking Description: The single-group assessment prohibits participant/outcomes masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-baseline Step Training (Experimental): Participants will be assessed before and after a 2-week baseline period, and again before and after a 2 week "protective step training period. Participants will also be assessed 2 months later at a follow-up visit.
  Interventions: Behavioral: Protective Step Training

INTERVENTIONS:
Behavioral: Protective Step Training — Participants will undergo 6, 1 hour visits (over the course of 2 weeks) where they will be exposed to repeated slips on a treadmill.

SUMMARY:
The primary purpose of this project is to determine the preliminary effectiveness of protective step training to improve balance and reduce falls in people with Parkinson's disease (PD) and postural disturbances. A secondary purpose is to understand which baseline patient characteristics predict responsiveness to treatment. By informing 1) the effectiveness of a promising rehabilitative intervention, and 2) the selection of the participants that will be most responsive to treatment, these data may enhance clinicians' ability to treat balance disturbances in people with PD. Importantly, protective step training, described in this proposal, can be quickly deployed in the clinic at minimal cost. Therefore, if shown to be effective via this and subsequent trials, this approach can be easily integrated into care, immediately impacting a large number of people with PD.

DETAILED DESCRIPTION:
This project contains 3 aims: Aims 1 and 2 address the primary goal of this project: Determining the effectiveness of protective step training. Aim 1 will test whether perturbation training can improve protective stepping in people with PD with postural dysfunction. Aim 2 will test whether improvements are retained over 2 months and generalize to untrained perturbation tasks (which may be important for real world situations). Importantly, investigators will also gather exploratory data regarding the effect of perturbation training on falls. Aim 3 addresses the secondary goal of this project: Determining for whom protective step training is most beneficial. Aim 3 will relate behavioral factors and neuroimaging outcomes to the magnitude of improvement in protective stepping. All aims will be tested in people with PD who have postural disturbances.

To complete these aims, participants will undergo 12 visits to the laboratory over the course of about 5 months. These will include 6 "training visits" over the course of 2 weeks, surrounded by 6 "assessment" visits before and after the training. During assessment visits, investigators will assess the ability to step quickly in response to a loss of balance (e.g. a slip), as well as thinking assessments and, if eligible, investigators will complete an MRI. During training visits, investigators will train the ability to step quickly in response to a slip.

In this study, participants will serve as their own controls. As such, there is no randomization to multiple groups.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist diagnosed PD
* Postural Instability / Gait Dysfunction (PIGD)
* Ability to stand unaided for 5 minutes

Exclusion Criteria:

* non-PD related neurological pathology
* orthopedic impairments affecting balance

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Stepping performance, measured as Margin of Stability (MOS) | Change across baseline period (2 weeks), compared to change across intervention period (2 weeks)
  MOS: Distance between the extrapolated center of mass and base of support at first foot contact after the slip

SECONDARY OUTCOMES:
Stepping performance, measured as First Step Length | Change across baseline period (2 weeks), compared to change across intervention period (2 weeks)
  Step Length: Length of the first step after the slip
Stepping performance, measured as First Step Latency | Change across baseline period (2 weeks), compared to change across intervention period (2 weeks)
  Step Latency: Time taken to lift the foot off the ground after the slip start
Cognition, measured as the total score on the "SCales for Outcomes in PArkinson's disease-COGnition" (SCOPA-COG) | Baseline
  SCOPA-COG: This scale characterizes cognitive capacity of several domains, and was developed specifically for people with PD. Range: 0-43 (higher score reflects better cognitive capacity). Subscales/domains are calculated, and the *total* score is calculated as the sum of each subscale.
Structural brain connectivity between the cortex (supplementary motor area), and basal ganglia (striatum) | Baseline
  Diffusion Tensor Imaging data (collected via MRI), will be collected and analyzed to characterize the structural connectivity specifically between the cortex and basal ganglia.

OTHER OUTCOMES:
Retention of stepping improvement (measured as Margin of Stability; MOS) over 2 months | Change in MOS score from Baseline to Follow-up (10 weeks between collections)
  Characterization of whether MOS changes observed over training period are retained at follow-up.
Generalization of stepping improvement (measured as Margin of Stability; MOS) | Change in MOS score from Baseline 2 to Post (2 weeks between collections)
  Characterize whether training impacts MOS of an untrained reactive stepping task
Fall frequency | Change in the number of falls during baseline (2 months) and follow-up (2 months) periods.
  Number of falls will be recorded via fall calendar in the 2 month period prior to training (baseline) and the 2 month period following training (post)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Peterson, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of the primary investigator and backup contact, noted above.

REFERENCES:
- [Derived] Monaghan AS, Hooyman A, Dibble LE, Mehta SH, Peterson DS. Stability Changes in Fall-Prone Individuals With Parkinson Disease Following Reactive Step Training. J Neurol Phys Ther. 2024 Jan 1;48(1):46-53. doi: 10.1097/NPT.0000000000000442. Epub 2023 Jun 1. PMID 37259190